CLINICAL TRIAL: NCT07040540
Title: The Effect of Intradermal Methylene Blue Application on Hemodynamic Stability Under General Anesthesia in Breast Surgery: A Prospective Observational Study
Brief Title: Hemodynamic Effects of Intradermal Methylene Blue During Breast Surgery Under General Anesthesia
Status: Completed | Type: Observational
Sponsor: Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Mustafa Kemal ŞAHİN, M.D, Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital
Other Study IDs: 2025-06/85
Record Dates: First submitted 2025-06-19; First posted 2025-06-27 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Breast Surgery; Sentinel Lymph Node Biopsy; Methylene Blue; Hemodynamic Stability; Intraoperative Hypotension
MeSH Terms: conditions — Breast Neoplasms | interventions — Methylene Blue; Coloring Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Methylene Blue Group: Patients undergoing elective breast surgery who receive an intradermal injection of 5 mL of 1% methylene blue for sentinel lymph node mapping.
  Interventions: Procedure: Methylene Blue
- Control Group: Patients undergoing elective breast surgery (mastectomy, lumpectomy, etc.) who do not receive methylene blue or any other dye injection, serving as a baseline for hemodynamic stability under general anesthesia.
  Interventions: Other: Standard Surgical Care Without Dye

INTERVENTIONS:
Procedure: Methylene Blue — Intradermal injection of 5 mL of 1% methylene blue solution administered into the breast tissue for sentinel lymph node mapping during breast cancer surgery. The dye is used to identify the first lymph nodes draining from the tumor site.
  Groups: Methylene Blue Group
Other: Standard Surgical Care Without Dye — Patients undergo standard breast surgery (mastectomy or lumpectomy) without administration of methylene blue or any other lymphatic mapping agent. All other perioperative care follows institutional standard protocols.
  Groups: Control Group

SUMMARY:
This prospective observational study aims to evaluate the effects of intradermal methylene blue injection on intraoperative hemodynamic stability in patients undergoing breast surgery under general anesthesia. While methylene blue is commonly used for sentinel lymph node mapping, its potential systemic vasopressor effects remain unclear. To provide a comprehensive analysis, the study will compare patients receiving methylene blue with a control group of patients undergoing similar breast procedures without the use of any dye. Hemodynamic parameters such as blood pressure, heart rate, and oxygen saturation will be recorded and compared between the two groups to determine the specific impact of methylene blue on the incidence of intraoperative hypotension and the need for vasopressor support.

DETAILED DESCRIPTION:
Sentinel lymph node biopsy is a standard procedure in breast cancer surgery to assess lymphatic spread. Methylene blue is widely used as a dye for sentinel lymph node mapping due to its safety, practicality, and cost-effectiveness. However, recent studies have suggested that methylene blue may have systemic vasopressor effects, particularly when it enters the circulation, by inhibiting guanylate cyclase and blocking nitric oxide pathways. This mechanism has been utilized in the management of refractory hypotension in septic shock, but its intraoperative hemodynamic effects during breast surgery remain unclear.

This prospective observational study will be conducted at Dr. Abdurrahman Yurtaslan Training and Research Hospital, Department of Anesthesiology and Reanimation, between August 1, 2025, and February 1, 2026. The study population will consist of two distinct cohorts: the Methylene Blue Group and the Control Group. Adult patients (aged 18-70) scheduled for elective breast surgery (mastectomy, lumpectomy, or sentinel lymph node biopsy) will be included. The Methylene Blue Group will consist of patients who receive intradermal methylene blue for sentinel lymph node mapping, while the Control Group will consist of patients undergoing breast surgery where no methylene blue or other mapping dyes are administered. All patients will be informed and written consent will be obtained prior to surgery. The study is entirely observational, with no intervention or alteration in the standard clinical management of patients.

Demographic data (age, BMI, ASA score), comorbidities, anesthesia protocols, methylene blue dose and timing (for the study group), and intraoperative hemodynamic parameters (blood pressure, heart rate, oxygen saturation) will be recorded for all participants. The incidence of intraoperative hypotension (defined as MAP <65 mmHg or a decrease of more than 20% from baseline) and the need for vasopressor support will be analyzed and compared between the two groups. Hemodynamic data will be collected at baseline (before anesthesia induction), immediately before methylene blue administration (or at a corresponding surgical time point for the control group), and at 5, 10, 15, 30, and 60 minutes after administration/reference point, as well as at the end of surgery.

The primary aim of this study is to assess and compare the impact of intradermal methylene blue on intraoperative hemodynamic stability against a control group in patients undergoing breast surgery under general anesthesia. By including a control group of patients who do not receive the dye, the study aims to isolate the specific hemodynamic effects of methylene blue from the general physiological changes associated with anesthesia and surgical stress. The results are expected to provide valuable information regarding the safety and potential vasopressor benefits of methylene blue in this context, helping anesthesia and surgical teams anticipate and manage possible hemodynamic changes during surgery. The findings may also contribute to the development of evidence-based protocols for the use of methylene blue in breast cancer surgery and guide future research in this area.

ELIGIBILITY:
Inclusion Criteria:

Female patients aged 18 to 70 years. Scheduled for elective breast surgery (mastectomy, lumpectomy, or sentinel lymph node biopsy).

For the study group: Planned use of intradermal methylene blue. For the control group: Breast surgery without the use of methylene blue. Provided written informed consent.

Exclusion Criteria:

Known allergy or hypersensitivity to methylene blue or other dyes Presence of severe cardiovascular disease Pregnancy Incomplete or missing data records

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Study Population: The study population consists of adult female patients, aged 18 to 70 years, who are scheduled for elective breast surgery at Dr. Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital. This population includes two distinct cohorts: (1) patients undergoing procedures that require sentinel lymph node mapping using intradermal methylene blue injection (such as breast-conserving surgery or mastectomy with SLNB), and (2) patients undergoing breast surgery (such as mastectomy or lumpectomy) where no methylene blue or other mapping dyes are administered, serving as the control group. All participants are selected from patients receiving general anesthesia and managed according to standard clinical protocols.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2026-01-10 (Actual)

PRIMARY OUTCOMES:
Comparison of Intraoperative Hemodynamic Stability Between Methylene Blue and Control Groups | From the induction of anesthesia until the end of the surgical procedure (approximately 1 to 3 hours per patient).
  The primary outcome is to compare the incidence of intraoperative hypotension (defined as a Mean Arterial Pressure <65 mmHg or a >20% decrease from baseline) and the total requirement for vasopressor administration (e.g., ephedrine, phenylephrine) between patients receiving intradermal methylene blue and the control group.

SECONDARY OUTCOMES:
Mean Arterial Pressure (MAP) and Heart Rate (HR) Trends | At specific intervals: Baseline, pre-injection, and 5, 10, 15, 30, 60 minutes after methylene blue administration or the corresponding surgical reference point.
  Comparison of the mean values of MAP and HR at specific intervals (baseline, pre-injection, and 5, 10, 15, 30, 60 minutes post-injection/reference point) between the two groups to identify the systemic vasopressor effect of methylene blue.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Kemal Şahin, Principal Investigator — Dr. Abdurrahman Yurtaslan Training and Research Hospital, University of Health Sciences
Locations (1):
- Dr. Abdurrahman Yurtaslan Ankara Oncology Education and Research Hospital Clinic of Anesthesiology and Rea, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Veronesi U, Paganelli G, Viale G, Galimberti V, Luini A, Zurrida S, Robertson C, Sacchini V, Veronesi P, Orvieto E, De Cicco C, Intra M, Tosi G, Scarpa D. Sentinel lymph node biopsy and axillary dissection in breast cancer: results in a large series. J Natl Cancer Inst. 1999 Feb 17;91(4):368-73. doi: 10.1093/jnci/91.4.368. PMID 10050871
- [Background] Kirov MY, Evgenov OV, Evgenov NV, Egorina EM, Sovershaev MA, Sveinbjornsson B, Nedashkovsky EV, Bjertnaes LJ. Infusion of methylene blue in human septic shock: a pilot, randomized, controlled study. Crit Care Med. 2001 Oct;29(10):1860-7. doi: 10.1097/00003246-200110000-00002. PMID 11588440
- [Background] Memis D, Karamanlioglu B, Yuksel M, Gemlik I, Pamukcu Z. The influence of methylene blue infusion on cytokine levels during severe sepsis. Anaesth Intensive Care. 2002 Dec;30(6):755-62. doi: 10.1177/0310057X0203000606. PMID 12500513